CLINICAL TRIAL: NCT02183688
Title: A Double-blind, Randomized, Placebo-controlled Clinical Trial to Confirm the Rationale of the ASA + Paracetamol + Caffeine Combination Compared With ASA + Paracetamol as Well as ASA, Paracetamol, and Caffeine in Headache Patients
Brief Title: Acetylsalicylic Acid (ASA) + Paracetamol + Caffeine Combination Compared With ASA + Paracetamol as Well as ASA, Paracetamol, and Caffeine in Headache Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 155.8
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Aspirin; Acetaminophen; Caffeine

ARMS (6):
- ASA + paracetamol + caffeine (Experimental)
  Interventions: Drug: Low dose ASA; Drug: Low dose paracetamol; Drug: Caffeine
- ASA + paracetamol (Active Comparator)
  Interventions: Drug: Low dose ASA; Drug: Low dose paracetamol
- ASA (Active Comparator)
  Interventions: Drug: High dose ASA
- Paracetamol (Active Comparator)
  Interventions: Drug: High dose paracetamol
- Caffeine (Active Comparator)
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose ASA
  Arms: ASA + paracetamol; ASA + paracetamol + caffeine
Drug: High dose ASA
  Arms: ASA
Drug: Low dose paracetamol
  Arms: ASA + paracetamol; ASA + paracetamol + caffeine
Drug: High dose paracetamol
  Arms: Paracetamol
Drug: Caffeine
  Arms: ASA + paracetamol + caffeine; Caffeine
Drug: Placebo
  Arms: Placebo

SUMMARY:
To confirm the combination rationale for the combination of ASA + paracetamol + caffeine compared with the combination of ASA + paracetamol and the individual substances ASA, paracetamol, caffeine, and placebo administered orally to headache patients for two headache episodes

ELIGIBILITY:
Inclusion Criteria:

1. Female or male out-patients aged between 18 and 65 years
2. Diagnosis: Headache

   1. Tension type headache according to international headache society (IHS) Headache Classification 2.1 (2.1.1 and 2.1.2) and/or
   2. Migraine according to IHS Headache Classification 1.1, 1.2.1 or
   3. Either a) or b), but cannot be distinctly classified
3. The patient normally treats his/her headache successfully with non-prescription analgesics
4. He/She has been suffering from headache for 12 months at least
5. The headache first occurred before the age of 50 years
6. During the previous three months, the patient has suffered from headache twice a month at least
7. Informed consent according to §§ 40, 41 of the german medicines act and Good Clinical Practice (GCP)
8. The patient seems likely to comply

Exclusion Criteria:

1. The patient treats his/her headache with prescription-only analgesics or migraine remedies
2. The patient requires higher single doses of non-prescription analgesics to treat his/her headache than indicated in the patient information leaflet (e.g. more than 2 tablets of Thomapyrin tablets)
3. The patient normally treats his/her headache with non-prescription analgesics in effervescent tablet form
4. The patient normally takes his/her non-prescription analgesics immediately at the onset of the first signs of a headache episode
5. Headache occurs on more than 10 days per month
6. The typical, untreated headache normally lasts less than 4 hours without treatment
7. Women with a close association between the occurrence of headache and menstruation (menstrual migraine)
8. Concomitant treatment with prescription-only and/or non-prescription analgesics
9. Previous or concomitant treatment with antidepressants or antipsychotic medicines (previous treatment = within the previous 4 weeks)
10. Previous or concomitant treatment with anti-rheumatic or anti-inflammatory drugs that may influence the headache symptoms (previous treatment = within the previous 4 days)
11. Treatment of concomitant illnesses with drugs containing ASA (above a daily dose of 100 mg per day), paracetamol or caffeine (e.g. for feverish common cold, etc.)
12. Migraine prophylaxis or administration of drugs, indicated for any other reasons that influence headache symptoms, e.g.

    Propanolol, Metoprolol, Flunarizine, Cyclandelate, Valproic acid, Serotonin antagonists (pizotifen, methysergide, lisuride), Ergotamine, Dihydroergotamine, Benzodiazepines, Magnesium, Monoamine oxidase inhibitors
13. Concomitant treatments with anti-emetics
14. Drug abuse connected with the headache (defined as the administration of analgesics or other drugs for the treatment of acute headache on more than 10 days per month)
15. Alcohol or drug abuse as defined by diagnostic and statistical manual of mental disorders (DSM-IV)
16. Pregnancy and lactation
17. Gastrointestinal ulcers
18. Pathologically increased bleeding tendency
19. Glucose-6-phosphate dehydrogenase deficiency
20. Hypersensitivity to paracetamol, caffeine, ASA, salicylates, and other anti-inflammatory/anti-rheumatic agents or other allergenic substances that are relevant to the clinical trial
21. Bronchial asthma
22. Concomitant treatment with anticoagulants (e.g. coumarin derivates, heparin)
23. Clinically relevant chronic or recurrent gastrointestinal symptoms
24. Clinically relevant liver disorders
25. Clinically relevant pre-existing renal damage
26. Gilbert's syndrome
27. Not successfully treated hyperthyroidism
28. Simultaneous participation in another clinical trial
29. Participation in another clinical trial within 4 weeks of entering this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1889 (Actual)
Dates: Start 1998-09; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Calculated time to 50% pain relief, based on the pain intensity evaluated on a visual analogue scale (VAS) | 30 min., 1, 2, 3 and 4 hours after administration of the study medication

SECONDARY OUTCOMES:
Percentage of patients with 50 % pain relief, evaluated on a VAS | At least 2 hours after administration of the study medication
Percentage of patients with 50 % pain relief, evaluated on a VAS | At least 30 min., 1, 3, and 4 hours after administration of the study medication
Pain intensity, evaluated on a VAS | 30 min., 1, 2, 3 and 4 hours after administration of the study medication
Ratio of weighted sum of pain intensity difference scores to maximum achievable sum of pain intensity differences (%SPIDweighted), evaluated on a VAS | Up to the end of the study
Extent of impairment of daily activities, evaluated on a 4-grade verbal scale (VRS) | Before, 30 min., 1, 2, 3 and 4 hours after administration of study drug
Duration of headache | Up to 48 hours after onset of each headache episode
Global assessment of efficacy by the patient, evaluated on a 4-grade VRS | Within 12 hours after study drug administration
Global assessment of tolerability by the patient, evaluated on a 4-grade VRS | Within 12 hours after study drug administration
Number of patients with adverse events | Up to the end of the study
Global assessment of tolerability by the investigator, evaluated on a 4-grade VRS | After each administration of study drug during the treatment phase